CLINICAL TRIAL: NCT02455661
Title: Femoral Closure Versus Radial Compression Devices Related to Percutaneous Coronary Interventions Study
Acronym: FERARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Sub-PI, Universitätsmedizin Mannheim
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-560N-MA
Record Dates: First submitted 2015-05-14; First posted 2015-05-28 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Arterial Closure Device; Percutaneous Coronary Intervention (PCI); Access Site Bleeding; Adverse Cardiac Events
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Radial closure by TR-Band.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Radial PCI with TR Band (TM) (Experimental): Patients with a PCI using the radial approach and the above radial compression device.
  Interventions: Device: TR Band (TM)
- Femoral PCI with AngioSeal device (Active Comparator): Patients with a PCI using the femoral approach and the above femoral vascular closure device.
  Interventions: Device: AngioSeal
- Femoral PCI with StarClose device (Active Comparator)
  Interventions: Device: StarClose

INTERVENTIONS:
Device: TR Band (TM)
  Arms: Radial PCI with TR Band (TM)
Device: AngioSeal
  Arms: Femoral PCI with AngioSeal device
Device: StarClose
  Arms: Femoral PCI with StarClose device

SUMMARY:
FERARI is a single centre observational study comparing patients undergoing PCI either using radial compression devices or femoral closure devices at the corresponding access site.

First primary outcomes consist of the occurrence of vascular complications at the arterial access site including major bleedings as defined by common classification systems

Second primary outcomes consist of the occurrence of adverse cardiac events including all-cause mortality, target lesion and vessel revascularization (TLR and TVR) during 30 days and 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent about the study
* Elective PCI with following indications:

Stable coronary artery disease, proven myocardial ischemia; cardiac arrhythmia; syncope; Unstable AP defined as NSTEMI but without cardiac troponin elevation; NSTEMI; STEMI

* patient eligible for coronary angiography and both radial and femoral PCI
* requirement of using a vascular closure device (without contraindications)

Exclusion Criteria:

* inability to understand and sign the informed consent term
* pregnancy
* less 18 years of age
* single diagnostic coronary angiography
* active or high bleeding risk (thrombocytopenia <50,000/µl)
* femoral approach and PCI without using a vascular closure device
* other conditions hampering involvement in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Vascular complications at the arterial access site | 30 days
  Occurrence of vascular complications at the arterial access site including major bleedings as defined by common classification systems
Adverse cardiac events | 30 days
  Occurrence of adverse cardiac events including all-cause mortality, target lesion and vessel revascularization (TLR and TVR).
Adverse cardiac events | 12 months
  Occurrence of adverse cardiac events including all-cause mortality, target lesion and vessel revascularization (TLR and TVR).

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Medicine, University Medical Centre Mannheim, Mannheim, Germany

REFERENCES:
- [Derived] Sartorius B, Behnes M, Unsal M, Hoffmann U, Lang S, Mashayekhi K, Borggrefe M, Akin I. Arterial access-site complications after use of a vascular closure device related to puncture height. BMC Cardiovasc Disord. 2017 Feb 16;17(1):64. doi: 10.1186/s12872-017-0484-7. PMID 28209184
- [Derived] Fastner C, Behnes M, Unsal M, El-Battrawy I, Ansari U, Mashayekhi K, Hoffmann U, Lang S, Kuschyk J, Borggrefe M, Akin I. Clinical outcomes of femoral closure compared to radial compression devices following percutaneous coronary intervention: the FERARI study. Heart Vessels. 2017 May;32(5):520-530. doi: 10.1007/s00380-016-0901-3. Epub 2016 Nov 1. PMID 27803954